CLINICAL TRIAL: NCT01387516
Title: Motivation and Skills for Detained Teen Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Responsible Party: Principal Investigator, Lynda Stein, Ph.D., Professor, University of Rhode Island
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: R01DA020731 (NIH)
Record Dates: First submitted 2011-05-25; First posted 2011-07-04 (Estimated); Results first posted 2020-04-20 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Motivational Intervention; Nicotine Anonymous; Cognitive Behavior Therapy; Relaxation Therapy
Keywords: nicotine; juveniles; detention
MeSH Terms: interventions — Motivational Interviewing; Relaxation Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This clinical trial uses a 2 x 2 between groups factorial design to investigate Motivational Interviewing versus Relaxation Therapy and Cognitive Behavior Therapy versus Self-Help Programming.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Motivational Intervention (Experimental): Motivational Interviewing (MI) will be a 60-90 minutes individual session.The focus is on establishing rapport and building motivation. The counselor explores youth's reasons for entering treatment, prior treatment experience, previous attempts to change use, possible goals for treatment, substance effect expectancy, and perceptions of self-efficacy. A personalized feedback report outlines assessment results, highlights any problems or concerns related to cigarette use expressed by teen, and compares tobacco use levels with national norms for same age and gender peers.
  Interventions: Behavioral: Motivational Intervention
- Relaxation Intervention (Active Comparator): The Relaxation Therapy intervention is a 60-90 minute individual session. The session encompasses several techniques, including Progressive Muscle Relaxation and Visualization-Imagination, and as a whole is really a meditation protocol.
  Interventions: Behavioral: Relaxation Therapy
- Cognitive Behavioral Therapy (Experimental): The Cognitive Behavioral Therapy (CBT) Intervention is administered during two 90 minute group sessions. The focus is on the interrelationship between thoughts, feelings, and behaviors. It is used to address specific deficits, such as improving problem solving skills and developing social supports, and behaviors such as substance abuse and smoking.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Self-Help Programming (Active Comparator): Self Help intervention is administered during two 90 minute group sessions. The intervention modules are based on the principles of Nicotine Anonymous (NicA), to provide those who use nicotine but wants a nicotine-free life, with a community of people that has also experienced nicotine addiction and strives to be nicotine free. Elements incorporated in this intervention include the 12 Steps and the NicA "tools" (i.e., meetings, phone list, literature, sponsorship, and service) to facilitate and maintain abstinence from nicotine.
  Interventions: Behavioral: Self-Help Programming

INTERVENTIONS:
Behavioral: Motivational Intervention — The MI session will be 60-90 minutes in length.The focus is on establishing rapport and building motivation. The counselor explores teen's reasons for entering treatment, prior treatment experience, previous attempts to change use, possible goals for treatment, substance effect expectancies, and perceptions of self-efficacy.A personalized feedback report outlines assessment results, highlights any problems or concerns related to cigarette use expressed by teen, and compares tobacco use levels with national norms for same age and gender peers.
  Other Names: Motivational Enhancement Therapy
  Arms: Motivational Intervention
Behavioral: Relaxation Therapy — The Relaxation Therapy intervention encompasses several techniques, including Progressive Muscle Relaxation and Visualization-Imagination, and meditation to reduce stress; which may lead to substance use.
  Arms: Relaxation Intervention
Behavioral: Cognitive Behavioral Therapy — The Cognitive-Behavioral Therapy (CBT) Intervention focuses on the interrelationship between thoughts, feelings, and behaviors. It addresses specific deficits, such as improving problem solving skills and developing social supports, and behaviors such as substance abuse and smoking.
  Arms: Cognitive Behavioral Therapy
Behavioral: Self-Help Programming — The Self-Help Programming intervention combines elements of Nicotine anonymous (NicA) to provide someone who uses nicotine but wants a nicotine-free life, with a community of people that has also experienced nicotine addiction and strives to be nicotine free. It incorporate the 12 Steps and the NicA "tools" (i.e., meetings, phone list, literature, sponsorship, and service) to facilitate and maintain abstinence from nicotine.
  Other Names: Nicotine Anonymous
  Arms: Self-Help Programming

SUMMARY:
The long-term objective of this research is to increase the investigators understanding of effective smoking interventions for understudied adolescents at high risk for continued smoking into adulthood.

This randomized clinical trial uses a 2 x 2 between groups design to investigate Motivational Interviewing (MI) versus Relaxation Therapy (RT), and Cognitive Behavior Therapy (CBT) versus Self-Help Programming (SHP). Treatments are provided during brief stay in detention and adolescents are followed after release. The investigators seek to increase quit rates post-release, and the investigators will examine the moderating and mediating effects of motivation, anger, and self-efficacy. The investigators will study main effects for treatment as well as whether the combination of MI/CBT is more effective than other treatments in enhancing quit rates.

Frequently, treatment for smoking cessation is unavailable to youths in the juvenile justice system, and when treatment is available, it may be provided using untested therapies. This study extends previous research by rigorously evaluating smoking cessation interventions specifically for teens at highest risk for continued smoking in adulthood. The investigators will examine processes contributing to the efficacy of treatments. The development of effective smoking interventions for juvenile detainees has the potential to reduce a significant public health concern in this undeserved and high-risk population.

DETAILED DESCRIPTION:
Research efforts to affect adolescent smoking cessation have not focused on detained teens. This is an opportune time to enhance interest in smoking cessation and subsequent quit rates. In addition, little is known about mechanisms of smoking cessation in adolescents, generally. The long-term objective of this research is to increase our understanding of effective smoking interventions for understudied adolescents at high risk for continued smoking into adulthood.

This Randomized Clinical Trial (RCT) uses a 2 x 2 between groups factorial design to investigate Motivational Interviewing (MI) versus Relaxation Therapy (RT), and Cognitive Behavior Therapy (CBT) versus Self-Help Programming (SHP). Treatments are provided during brief stay in detention and adolescents are followed after release. The investigators seek to increase quit rates post-release, and the investigators will examine the moderating and mediating effects of motivation, anger, and self-efficacy. The investigators will study main effects for treatment as well as whether the combination of MI/CBT is more effective than other treatments in enhancing quit rates.

Methodology-Adolescents ages 13-19, who have been detained at the Rhode Island Training School (RITS; ethnic breakdown: 32% Caucasian, 35% African American, 22% Latino, 5% Asian American, and 6% of other racial backgrounds),and approximately 10% of its residents are female. Adolescents will be eligible if: 1) they smoke an average of 1 cigarette or cigarillo per day 2) they have an estimated length of 4-7 weeks stay in detention.

All teens who meet the inclusion criteria will be initially introduced to the study by Rhode Island Training School (RITS) authorized personnel who will briefly explain the study. Youth will be approached in person at the facility and if interested in the study, project staff describes the purposes, procedures, and answers all questions the youth may have.It is also emphasized that to not participate will not result in any repercussions in terms of their detention to the facility.

In order to participate in the study, eligible teens will be required to read (or have read) and sign an informed consent/assent form. Teens not meeting screening criteria or who decline participation in the study will be thanked for their time. Teens who meet the inclusion criteria, but decline participation will be asked to fill out a brief, anonymous questionnaire containing demographic information and items concerning previous incarcerations. If they agree to do so, they will be asked to read and sign an informed consent/assent form. The purpose of this brief questionnaire is to allow us to determine if the sample of teens that agreed to participate is significantly different from those who declined.

After obtaining informed consent/assent, Youth complete the baseline assessment which takes approximately 105 minutes to complete. All information will be collected during an interview with a trained Research Assistant (RA), including an orientation to the project. These assessments are identical for all conditions and will occur within 24 hrs. of consent/assent at the RITS.

Contact information including; addresses, numbers, nicknames, employer info., and school info, driver's license numbers, case workers (CW), probation officers (PO), and two family or friends who would be able to locate them will be recorded.Locator information will include name, address, and phone number, relation to the teen.Youth will be asked to sign a letter addressed to their locators that explains that they are participating in a research project at the University of Rhode Island (URI) and that they have given permission for the locator to provide project staff with information to locate him/her.This letter provides no information about the nature of the project.Locators will be contacted only if all other attempts to reach the teen have failed.

Youth are then urn randomized to receive either one individual session of Motivational Interviewing (MI) or Relaxation Therapy (RT). To optimize our chances of establishing a causal relationship between the treatment conditions and differential treatment outcome urn randomization is be employed. For our purposes age (<16 vs. > 16),family history of smoking (none vs. first degree biological relatives), and childhood onset conduct disorder with aggressive symptoms (yes vs. no) will factor into the urn randomization procedure, making it more likely that groups will balance on these variables.

The MI session is 60-90 minutes in length, with focus on establishing rapport and building motivation. The counselor explores teen's reasons for entering treatment, prior treatment experience, previous attempts to change use, possible goals for treatment, substance effect expectancy, and perceptions of self-efficacy. A personalized feedback report outlines assessment results, highlights any problems or concerns related to cigarette use expressed by teen, and compares tobacco use levels with national norms for same age and gender peers.

The RT condition is designed to be comparable in time to the MI, thus participants in this condition will meet individually with a therapist for 60-90 minutes on one occasion. These sessions will focus on instruction in muscle relaxation and meditation, and youth will be given feedback and handouts on use of relaxation techniques. This relaxation training protocol has been used as a treatment condition in a number of Institutional Review Board (IRB) approved intervention studies.

After receiving one individualized treatment, youth are then randomized to one of two different group interventions.

Cognitive Behavioral Therapy (CBT) sessions will focus on training a variety of skills including problem solving, coping, refusal of tobacco, communication, identification of appropriate support networks, and developing a personal emergency plan for after release. Each of these two group sessions at 60-75 minutes in length.

Self-Help Programming (SHP) utilizes a Nicotine Anonymous (NicA) approach to group treatment. Therefore, the 12-step philosophy, tools and traditions of NicA, and what is gained by giving up nicotine are discussed along with tips for not smoking. Each of these two group sessions are 60-75 minutes in length.

A thirty minute Post-Individual Assessment (FFU1) occurs after the individual MI or RT session. A 45 minute Post-Group Assessment (FFU2) occurs at the end of the youth's last group session. These assessments are conducted by a Research Assistant (RA) blind to treatment assignment.These assessments tap retention of experimental treatment effects.Incentives include snacks and individual attention.

A RA will schedule a post-release three month follow up assessment prior to the youth's release from RITS. The assessment will vary depending on when the teen is released, however the assessment will take place 3 months after the release date for each teen. The remaining Follow up is six months post release and is scheduled by the RA conducting the previous session. Each follow-up assessments are approximately 60-90 minutes in length and will be conducted in person in a private office at the University of Rhode Island, by a trained RA. Assessments consist of questions regarding post-release behaviors such as previous charges, smoking, and self-efficacy, and will utilize the same measures used in the baseline assessment.

ELIGIBILITY:
Inclusion Criteria:

* 13-19 years old,
* smokes average of 1 cigarette or cigarillo per day
* in facility for at least 4 days.

Exclusion Criteria:

* non-smoker,
* not in facility long enough (i.e. 4 days).

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 314 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Stein, Ph.D., Principal Investigator — University of RI
Locations (1):
- Rhode Island Training School, Cranston, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 18 participants who were enrolled and completed the baseline assessment either withdrew or were lost prior to treatment assignment.
Groups:
- Motivational Intervention/Cognitive Behavioral Therapy: Motivational Intervention (MI) is one 60-90 minute individual session focusing on establishing rapport and building motivation. The counselor explores teen's reasons for entering treatment, prior treatment experience, previous attempts to change use, possible goals for treatment, substance effect expectancies, and perceptions of self-efficacy. This is followed by two 90 minute Cognitive Behavioral Therapy (CBT) group sessions focusing on the interrelationship between thoughts, feelings, and behaviors. It is used to address specific deficits, such as improving problem solving skills and developing social supports, and behaviors such as substance abuse and smoking.
- Motivational Interviewing/Self-Help Programming: Motivational Intervention (MI) is one 60-90 minute individual session focusing on establishing rapport and building motivation. The counselor explores teen's reasons for entering treatment, prior treatment experience, previous attempts to change use, possible goals for treatment, substance effect expectancies, and perceptions of self-efficacy. This is followed by two 90 minute group Self Help intervention sessions based on the principles of Nicotine Anonymous (NicA), to provide those who use nicotine but wants a nicotine-free life, with a community of people that has also experienced nicotine addiction and strives to be nicotine free. Elements incorporated in this intervention include the 12 Steps and the NicA "tools" (i.e., meetings, phone list, literature, sponsorship, and service) to facilitate and maintain abstinence from nicotine.
- Relaxation Intervention/Cognitive Behavioral Therapy: The Relaxation Therapy intervention one 60-90 minute individual session that encompasses several techniques, including Progressive Muscle Relaxation and Visualization-Imagination, and as a whole is really a meditation protocol. This is followed by two 90 minute Cognitive Behavioral Therapy (CBT) group sessions focusings on the interrelationship between thoughts, feelings, and behaviors. It is used to address specific deficits, such as improving problem solving skills and developing social supports, and behaviors such as substance abuse and smoking.
- Relaxation Intervention/Self-Help Programming: The Relaxation Therapy intervention is one 60-90 minute individual session that encompasses several techniques, including Progressive Muscle Relaxation and Visualization-Imagination, and as a whole is really a meditation protocol. This is followed by two 90 minute group sessions of Self Help intervention, based on the principles of Nicotine Anonymous (NicA), to provide those who use nicotine but wants a nicotine-free life, with a community of people that has also experienced nicotine addiction and strives to be nicotine free. Elements incorporated in this intervention include the 12 Steps and the NicA "tools" (i.e., meetings, phone list, literature, sponsorship, and service) to facilitate and maintain abstinence from nicotine.
Period: Overall Study
Arm/Group | Motivational Intervention/Cognitive Behavioral Therapy | Motivational Interviewing/Self-Help Programming | Relaxation Intervention/Cognitive Behavioral Therapy | Relaxation Intervention/Self-Help Programming
Started | 80 | 68 | 79 | 69
Completed | 75 | 63 | 75 | 65
Not Completed | 5 | 5 | 4 | 4
Not completed — Lost to Follow-up | 4 | 4 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Motivational Intervention/Cognitive Behavioral Therapy: Motivational Intervention (MI) is one 60-90 minute Individual session focused on establishing rapport and building motivation. Followed by two 90 minute Cognitive Behavioral Therapy (CBT) group sessions focused on the interrelationship between thoughts, feelings, and behaviors. It is used to address specific deficits, such as improving problem solving skills and developing social supports, and behaviors such as substance abuse and smoking.
- Motivational Intervention/Self-Help Programming: Motivational Intervention (MI) is one 60-90 minute Individual session focused on establishing rapport and building motivation. Followed by two 90 minute Self Help Intervention group sessions based on the principles of Nicotine Anonymous (NicA), to provide those who use nicotine but wants a nicotine-free life, with a community of people that has also experienced nicotine addiction and strives to be nicotine free.
- Relaxation Intervention/Cognitive Behavioral Therapy: The Relaxation Therapy intervention is one 60-90 minute individual session, encompassing Progressive Muscle Relaxation and Visualization-Imagination, and as a whole is really a meditation protocol. This is followed by two 90 minute Cognitive Behavioral Therapy (CBT) group sessions focused on the interrelationship between thoughts, feelings, and behaviors. It is used to address specific deficits, such as improving problem solving skills and developing social supports, and behaviors such as substance abuse and smoking.
- Relaxation Intervention/ Self-Help Programming: The Relaxation Therapy intervention is one 60-90 minute individual session, encompassing Progressive Muscle Relaxation and Visualization-Imagination, and as a whole is really a meditation protocol. This is followed by two 90 minute Self Help intervention group sessions based on the principles of Nicotine Anonymous (NicA), to provide those who use nicotine but wants a nicotine-free life, with a community of people that has also experienced nicotine addiction and strives to be nicotine free.
- Total: Total of all reporting groups
Arm/Group | Motivational Intervention/Cognitive Behavioral Therapy | Motivational Intervention/Self-Help Programming | Relaxation Intervention/Cognitive Behavioral Therapy | Relaxation Intervention/ Self-Help Programming | Total
Number analyzed (Participants) | 80 | 68 | 79 | 69 | 296
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.65 (1.07) | 16.83 (1.00) | 16.75 (1.13) | 16.46 (1.21) | 16.68 (1.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 8 | 17 | 11 | 52
  Male | 64 | 60 | 62 | 58 | 244
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 26 | 20 | 16 | 80
  Not Hispanic or Latino | 62 | 42 | 59 | 53 | 216
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 4 | 3 | 10
  Asian | 2 | 4 | 0 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 2 | 0 | 3
  Black or African American | 21 | 15 | 13 | 11 | 60
  White | 55 | 47 | 60 | 54 | 216
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cigarette Use, Average # of Cigarettes Per Smoking Day.
Description: Using a 60-day TLFB we collected the average number of cigarettes smoked per smoking day at 6-month follow-ups
Time Frame: 6 months post release
Population: Participants who received both individual (MI or RT) and group (CBT or SHP) treatment who received 6 month follow-up and who had at least one smoking day were included in this analysis. Non-smokers @ 6 month were excluded.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Motivational Interviewing/ Cognitive Behavioral Therapy: Motivational Intervention (MI) is one 60-90 minute Individual session focused on establishing rapport and building motivation. Followed by two 90 minute Cognitive Behavioral Therapy (CBT) group sessions focused on the interrelationship between thoughts, feelings, and behaviors. It is used to address specific deficits, such as improving problem solving skills and developing social supports, and behaviors such as substance abuse and smoking
- Motivational Interviewing/Self Help Programming: Motivational Intervention (MI) is one 60-90 minute Individual session focused on establishing rapport and building motivation. Followed by two 90 minute Self Help Intervention group sessions based on the principles of Nicotine Anonymous (NicA), to provide those who use nicotine but wants a nicotine-free life, with a community of people that has also experienced nicotine addiction and strives to be nicotine free.
- Relaxation Intervention/Self Help Programming: The Relaxation Therapy intervention is one 60-90 minute individual session, encompassing Progressive Muscle Relaxation and Visualization-Imagination, and as a whole is really a meditation protocol. This is followed by two 90 minute Self Help intervention group sessions based on the principles of Nicotine Anonymous (NicA), to provide those who use nicotine but wants a nicotine-free life, with a community of people that has also experienced nicotine addiction and strives to be nicotine free.
Arm/Group | Motivational Interviewing/ Cognitive Behavioral Therapy | Motivational Interviewing/Self Help Programming | Relaxation Intervention/Cognitive Behavioral Therapy | Relaxation Intervention/Self Help Programming
Number analyzed (Participants) | 67 | 55 | 58 | 54
days | 8.01 (6.52) | 8.87 (9.07) | 8.89 (7.29) | 7.55 (6.35)

2. Primary Outcome: Number of Subjects Who Were Verified Abstinent From Smoking Using CO Levels and Cotinine in the Saliva
Description: A smokelyzer and a saliva sample are used to get information on CO levels and cotinine in the saliva as biochemical markers for our research. These levels will determine if the participant is verified as being abstinent from smoking during the week before collection.
Time Frame: 6 months post release
Population: All participants that supplied biochemical markers. If a participant was lost at 3 month follow up; Baseline biochemical markers were included in analysis. When a participant was lost at 6 month follow up, 3 month biochemical markers were used in analysis. 1 participant in the RT/SHP arm never submitted biochemical markers and is not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interviewing/ Cognitive Behavioral Therapy | Motivational Interviewing/Self Help Programming | Relaxation Intervention/Cognitive Behavioral Therapy | Relaxation Intervention/Self Help Programming
Number analyzed (Participants) | 80 | 68 | 79 | 68
Participants | 15 | 15 | 18 | 15

3. Primary Outcome: American Thoracic Society Questionnaire (ATSQ)
Description: This validated 8 item measure assesses the frequency of experiencing several respiratory symptoms using a 5 point Likert scale from 1, never to 5, every day. The minimum score is 8 indicating no experience of respiratory symptoms and the maximum score is 40 which indicates a high frequency of experiencing respiratory symptoms.
Time Frame: 6 months post release
Population: Participants who received individual (MI or RT) and group treatment (CBT or SHP) and who also received a 6 month follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivational Interviewing/ Cognitive Behavioral Therapy | Motivational Interviewing/Self Help Programming | Relaxation Intervention/Cognitive Behavioral Therapy | Relaxation Intervention/Self Help Programming
Number analyzed (Participants) | 75 | 63 | 75 | 65
score on a scale | 16.11 (6.36) | 16.65 (6.83) | 15.26 (6.64) | 15.91 (6.53)

4. Primary Outcome: Percent Smoking Days
Description: Using a Time-Line Follow-back, we calculated percent smoking days for a 60 day period at 6-month follow-up. This is the percentage of smoking days a participant had out of possible smoking days (days for which the participant was not in a controlled environment where they did not have access to cigarettes).
Time Frame: 6 months post release
Population: Includes participants who received individual (MI or RT) and group (CBT or SHP) treatment who also had a 6 month follow up and access to cigarettes. Participants who spent all 90 days of this assessment period in a controlled environment where they did not have access to cigarettes were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: percentage of smoking days
Arm/Group | Motivational Interviewing/ Cognitive Behavioral Therapy | Motivational Interviewing/Self Help Programming | Relaxation Intervention/Cognitive Behavioral Therapy | Relaxation Intervention/Self Help Programming
Number analyzed (Participants) | 70 | 55 | 68 | 58
percentage of smoking days | 83.20 (32.53) | 87.34 (24.68) | 68.17 (38.75) | 81.62 (33.22)

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Motivational Intervention/Cognitive Behavioral Therapy | Motivational Interviewing/Self-Help Programming | Relaxation Intervention/Cognitive Behavioral Therapy | Relaxation Intervention/Self-Help Programming
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/68 | 0/79 | 1/69
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/68 | 0/79 | 0/69
Other Adverse Events (participants affected / at risk) | 0/80 | 0/68 | 0/79 | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes